CLINICAL TRIAL: NCT07289425
Title: The Effect of a Mobile Application Developed for Obese Children on Eating Attitudes, Eating Awareness, and Healthy Eating Self-Efficacy
Brief Title: Effect of a Mobile App for Obese Children on Eating Attitudes, Eating Awareness, and Healthy Eating Self-Efficacy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Nurcan Karamercimek, Master's Degree Student, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SCÜ-HMŞ-NK-01
Record Dates: First submitted 2025-11-15; First posted 2025-12-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Child Health
Keywords: Child health; obesity; eating behavior; mindful eating; self efficacy
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Preliminary information will be provided and consent will be obtained. The introductory information form, the eating attitude test for children, the eating awareness scale, and the healthy eating self-efficacy scale will be completed, and BMI calculations will be performed. These procedures will be repeated during the interim follow-up at the end of the first month and the final test at the end of the second month.
- working group (Experimental): Preliminary information will be provided and consent will be obtained. An introductory information form, a food attitude test for children, a food awareness scale, and a healthy eating self-efficacy scale will be completed, and BMI calculations will be performed. The mobile application will be introduced and downloaded to the parent's cell phone. An 8-week training program will be provided through the application. After one month, the scales will be reapplied during the interim follow-up and the BMI will be calculated. At the end of the second month, the scales will be reapplied for the final test and the BMI will be calculated.
  Interventions: Device: Childhood Obesity Mobile Application

INTERVENTIONS:
Device: Childhood Obesity Mobile Application — With the support of computer engineers and software experts, the logo, user interface, overall appearance, and control panel will be designed to suit the purpose and subject matter of the mobile application. The mobile application will be designed to be used on both Android and iOS-based smartphones and in environments without internet access. After developing the prototype of the mobile application, its usability will be tested. In this context, the testing process will first be carried out by researchers. Academic nurses (n=3) and outpatient clinic nurses (n=2) will evaluate the application using the Mobile Application Usability Scale. If any problems are identified in the application, they will be resolved and the necessary adjustments will be made.
  Arms: working group

SUMMARY:
This study aims to evaluate the effect of a mobile application developed for obese children on eating attitudes, eating awareness, and healthy eating self-efficacy. The application seeks to support children in developing healthy eating habits and to integrate nursing interventions with digital health technologies in combating obesity. Data will be collected through a researcher-developed Information Form and three validated scales: the Eating Attitude Test, the Eating Awareness Scale, and the Healthy Eating Self-Efficacy Scale, completed by both children and parents.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of a mobile application developed for obese children on their eating attitudes, eating awareness levels, and self-efficacy regarding healthy eating, with the aim of contributing to the integration of nursing interventions with digital health technologies in the fight against obesity. Increasing childhood obesity negatively affects not only physical health but also psychosocial development, necessitating multifaceted and sustainable interventions. In line with nurses' effective roles in health education and behaviour change, the application will be developed to support children in acquiring and maintaining healthy eating habits. Additionally, the integration of digital technologies into nursing care and their effectiveness in reaching families will be evaluated; this study will provide a unique contribution to this area, which is lacking in the literature.

The research data will be collected using the Information Form created by the researcher, the Healthy Eating Self-Efficacy Scale for Children, the Eating Attitude Test for Children, and the Eating Awareness Scale for Children.

A total of 18 questions comprising demographic characteristics of children and parents and their eating habits will be used to collect data for the study. In addition, the Eating Attitude Test, consisting of 26 items, will be used to assess eating behaviour and the risk of possible eating disorders in children aged 8-15 years. the 12-item Eating Awareness Scale to determine the degree to which children aged 8-11 are mindful or automatic while eating, and the 9-item Healthy Eating Self-Efficacy Scale to assess the perceived competence of children aged 8-10 in healthy eating. All forms and scales will be completed by children and parents.

ELIGIBILITY:
Inclusion Criteria:

* The child must be between 8 and 10 years old,
* The child must not have any chronic illnesses other than obesity,
* The child must be able to read and write in Turkish,
* The child must be able to use a mobile device,
* The child must not have a visual impairment,
* The parent must be willing to participate in the study,
* The parent must be able to read and write in Turkish,
* The parent or child must have a smartphone.

Exclusion Criteria:

* If they wish to withdraw from the study at any stage of the research,
* If they do not wish to use the mobile application at any stage of the research.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Eating Attitude Test for Children | At baseline, 4 weeks after the start of the intervention, and 8 weeks after the start of the intervention
  This scale is used to identify eating-related attitudes and behaviors among children aged 8-15. It consists of 26 items and evaluates general patterns indicating how children feel, think, and behave regarding eating, using a six-point Likert-type structure.
Eating Awareness Scale for Children | At baseline, 4 weeks after the start of the intervention, and 8 weeks after the start of the intervention
  This scale assesses the level of attention children aged 8-11 pay to food during eating behaviors and evaluates inattentive or automatic eating tendencies through its 12-item, two-dimension structure, using a four-point Likert-type format.

SECONDARY OUTCOMES:
Healthy Eating Self Efficacy Scale for Children | At baseline, 4 weeks after the start of the intervention, and 8 weeks after the start of the intervention
  This scale measures children's confidence in their ability to make healthy food choices and maintain healthy eating behaviors. It evaluates their perceived capability to engage in healthy eating practices and is designed for children aged 8-10. The scale consists of 9 items and uses a three-point Likert-type structure.
Body Mass Index | At baseline, 4 weeks after the start of the intervention, and 8 weeks after the start of the intervention
  Height and weight measurements will be used to calculate BMI (kg/m²) in participants.

CONTACTS AND LOCATIONS:
Overall Officials: İlknur Yıldız, Associate Professor, Study Chair — Sivas Cumhuriyet University, Faculty of Health Sciences
Locations (1):
- Sivas Cumhuriyet University, Sivas, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kocaadam-Bozkurt, B., Köksal, E., & Özalp Ateş, F. S. (2022). Mindful Eating Questionnaire for Children: Validation and reliability in Turkish children. Mindfulness, 13, 1469-1478. https://doi.org/10.1007/s12671-022-01889-5.
- [Background] Browne NT. Obesity and Children. Nurs Clin North Am. 2021 Dec;56(4):583-597. doi: 10.1016/j.cnur.2021.07.006. PMID 34749897
- [Background] Bozkurt O, Kocaadam-Bozkurt B, Koksal E, Ozalp Ates FS. Children's eating attitudes test (ChEAT): validation and reliability in Turkish children. J Eat Disord. 2023 Aug 31;11(1):93. doi: 10.1186/s40337-023-00811-1. PMID 37649120
- [Background] Kabasakal, E., Arslan, U. E., Üner, S., Konşuk Ünlü, H., Bilir, N., Yardım, M. S., Araz, Ö., Huang, T., & Özcebe, H. (2020). The Turkish validity and reliability study of the Healthy Eating Self-Efficacy Scale for Children. Türkiye Çocuk Hastalıkları Dergisi / Turkish Journal of Pediatric Disease, 14(1), 1-10. https://doi.org/10.12956/tchd.556078.